CLINICAL TRIAL: NCT04148170
Title: Recanalization of Congenital Nasolacrimal Duct Obstruction by Endodiathermy Probe and Intubation Versus Intubation Only
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Hassan Abdelbaky, Assistant Professor of Ophthalmology., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo118988
Record Dates: First submitted 2019-10-27; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Congenital Nasolacrimal Duct Obstruction
Keywords: Endodiathermy Probe and Intubation Versus Intubation Only

STUDY DESIGN:
Intervention Model Description: Group (I): 80 eyes of children suffer from congenital nasolacrimal duct obstruction will have probing with metal probe and then intubation with bicanlicular silicon tube.
  Group (II): 80 eyes of children suffer from congenital nasolacrimal duct obstruction will have probing with endodiathermy probe and then intubation with bicanlicular silicon tube.
Who Masked: Participant
Masking Description: all will be know the surgical procedure but participant will know only that he will be treated but cant understand type of procedure done
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic intubation (Active Comparator): children suffer from congenital nasolacrimal duct obstruction will have probing with metal probe and then intubation with bicanlicular silicon tube.
  Interventions: Procedure: Endodiathermy Probe and Intubation Versus Intubation
- endodiathermy probe (Active Comparator): children suffer from congenital nasolacrimal duct obstruction will have probing with endodiathermy probe and then intubation with bicanlicular silicon tube
  Interventions: Procedure: Endodiathermy Probe and Intubation Versus Intubation

INTERVENTIONS:
Procedure: Endodiathermy Probe and Intubation Versus Intubation — children suffer from congenital nasolacrimal duct obstruction will have probing with endodiathermy probe and then intubation with bicanlicular silicon tube

SUMMARY:
The purpose of the current work is to assess the efficiency and success rate of endodiathermy probe followed by intubation in children more than 2 years compared to the success rate of intubation (as a standard method) which varies from 75% to 85% in several studies

DETAILED DESCRIPTION:
The study will be conducted on children above 2 year and will be divided randomly into two groups:

Group (I): 80 eyes of children suffer from congenital nasolacrimal duct obstruction will have probing with metal probe and then intubation with bicanlicular silicon tube.

Group (II): 80 eyes of children suffer from congenital nasolacrimal duct obstruction will have probing with endodiathermy probe and then intubation with bicanlicular silicon tube

ELIGIBILITY:
Inclusion Criteria:

1. Children in the age group above 2 years old
2. No history of previous probing.
3. No history of previous intubation.
4. Children with no any other association or congenital anomalies cause watery eye.
5. children suffer from congenital nasolacrimal duct obstruction.

Exclusion Criteria:

1. children less than 2 years old.
2. previous probing.
3. previous intubation.
4. children with any other congenital anomalies as congenital ectropion , congenital entropion
5. children suffer from any upper lacrimal anomalies as obstruction or stenosis.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
recanalization of nasolacrimal duct | 6 months
  compare the efficiency of endodiathermy probe followed by intubation versus probing with metal probe followed by intubation by
  1. epiphora (overflow of tears onto the face)
  2. increase tear film meniscus ( more than 1mm in height)
  3. mucous discharge
  4. Fluorescein disappearance test (Normally, little or no dye remains after 5 minutes. Prolonged retention is indicative of inadequate lacrimal drainage)

SECONDARY OUTCOMES:
complication | 6 months
  Record any complication in two procedures as tube migration, tube extrusion, infection or need for additional procedure.

CONTACTS AND LOCATIONS:
Overall Officials: tamer gawdat, professor, Principal Investigator — professor of ophthalmology cairo university
Locations (1):
- Abo El Resh Pedriatric Hospital Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after finishiny my research can share my data
Supporting Information: Study Protocol, ICF
Time Frame: 1 year untill 1 year and 6 months
Access Criteria: after finish my study

REFERENCES:
- [Result] Suranagi PV, Poornima MS; Smruthi; Banagar B. Regarding a novel technique to recanalize the nasolacrimal duct with endodiathermy bipolar probe. Indian J Ophthalmol. 2014 Sep;62(9):971. doi: 10.4103/0301-4738.143956. No abstract available. PMID 25370408